CLINICAL TRIAL: NCT01322334
Title: A Single Blinded Prospective Randomized Controlled Trial to Investigate Whether Singing Exercises Can Improve Symptoms of Snoring and Sleep Apnea
Brief Title: Singing Exercises to Improve Symptoms of Snoring and Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Malcolm Hilton, Consultant Otolaryngologist and Clinical Lecturer, Royal Devon & Exeter hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hil2003/SE
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-03

CONDITIONS: Snoring; Upper Airway Resistance Syndrome; Obstructive Sleep Apnea
Keywords: Snoring; Sleep apnea; Pharyngeal muscle tone
MeSH Terms: conditions — Snoring; Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Singing exercises (Experimental)
  Interventions: Behavioral: Singing exercises

INTERVENTIONS:
Behavioral: Singing exercises — A 3 month self-guided treatment based on a specially designed 3CD box set, which patient performed every day ('Singing for Snorers': UK)

SUMMARY:
Upper airway resistance during sleep can present with a range of symptoms from simple snoring (SS) through to severe obstructive sleep apnea (OSA). Pharyngeal narrowing or collapse leads to reduction or cessation in airflow during sleep, and is associated with loud snoring.

The investigators hypothesized that regular singing exercises could strengthen pharyngeal muscles and/or increase their resting tone, and lead to an improvement of symptoms and thus quality of life in patients with all forms of snoring.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years old or over
* history of simple snoring or sleep apnoea with RDI 10-40

Exclusion Criteria:

* severe sleep apnoea RDI >40
* morbid obesity BMI > 40
* unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2005-11; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Epworth sleepiness scale | Entry to study (day one), and after 3 months of intervention

SECONDARY OUTCOMES:
Loudness of snoring | Entry to study (day one), and 3 months after intervention
  Visual analogue scale rating
Frequency of snoring | Entry to study (day one), and 3 months after intervention
  Visual analogue scale rating
SF-36 quality of life assessment tool | Entry to study (day one), and 3 months after intervention
Compliance with exercises | After 3 months of intervention
  Applied only to intervention group. Rated on visual analogue scale of 100mm from 'never' to 'every day'

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm P Hilton, BMBCh FRCS, Principal Investigator — Royal Devon and Exeter NHS Foundation Trust
Locations (1):
- Royal Devon & Exeter NHS Foundation Trust, Exeter, United Kingdom